CLINICAL TRIAL: NCT05972421
Title: Impact of Proactive Outreach on Enrollment in and Utilization of the Flex Nutrition Program for Patients With Food Insecurity and Nutritionally Dependent Chronic Health Conditions
Brief Title: Enrollment in and Utilization of the Flex Nutrition Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sarah A. Matathia, MD, MPH, Associate Medical Director of Primary Care Equity, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P002954
Record Dates: First submitted 2023-07-14; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Food Insecurity; Vulnerable Populations; Nutrition, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Proactive Outreach (Experimental): Patients will receive a mailed letter as well as proactive outreach by phone. The objective of the letter and phone outreach is to describe the Flex Nutrition Program and offer enrollment.
  Letters will be written in the primary language spoken by the patient. The letter will contain a call back phone number as well as a primary email contact. Patients will be provided with the phone number of Interpreter Services to utilize if needed.
  1 week following the mailing of the letter, patients will receive 3 phone calls within 10 business days, occurring at different times of day. Patients will be provided a call back number. Phone calls will be made to patients in their primary languages, with the use of Interpreters as needed.
  Interventions: Other: High Intensity Proactive Outreach
- Low Intensity Proactive Outreach (Experimental): Patients will receive a mailed letter. The objective of the letter is to describe the Flex Nutrition Program and offer enrollment.
  Letters will be written in the primary language spoken by the patient. The letter will contain a call back phone number as well as a primary email contact. Patients will be provided with the phone number of Interpreter Services to utilize if needed.
  Interventions: Other: Low Intensity Proactive Outreach
- No Outreach; Usual Care (No Intervention): Patients will not receive any proactive outreach and will serve as a comparison group. These patients may be referred to the Flex Nutrition Program through their Care Managers.

INTERVENTIONS:
Other: High Intensity Proactive Outreach — phone calls + mailed letter to eligible patients to describe and offer enrollment into the FLEX Nutrition Program
  Arms: High Intensity Proactive Outreach
Other: Low Intensity Proactive Outreach — mailed letter to eligible patients to describe and offer enrollment into the FLEX Nutrition Program
  Arms: Low Intensity Proactive Outreach

SUMMARY:
The goal of this clinical trial is to learn about the impact of proactive outreach on enrollment into and utilization of the Flexible Services Nutrition Program. The Flexible Services Nutrition Program increases access to healthy foods for patients with Medicaid ACO insurance, food insecurity and nutritionally dependent chronic health conditions.

The main questions the study aims to answer are:

* Does proactive outreach to eligible patients increase enrollment into the Medicaid ACO FLEX Nutrition Program, compared to usual care?
* Does high intensity outreach (letter +phone calls) increase enrollment more than low intensity outreach (letter only)?

The investigators will also conduct exploratory analyses to evaluate if proactive outreach has an effect on healthcare utilization (ED visits, unplanned hospitalizations, and outpatient no-show rate) and health outcomes (BMI for patients with overweight/obesity, a1c for patients with impaired fasting glucose/Diabetes, Blood Pressure for patients with Hypertension).

DETAILED DESCRIPTION:
The Medicaid ACO Flexible Services Program is a pilot that allocates state funding to address certain health-related social needs, in the domains of food and housing, with the goal of improving health outcomes and reducing the total cost of health care for members. The Flex Nutrition Program specifically allows members with a health needs-based criteria (such as a complex physical health need, repeated Emergency Department use or a high-risk pregnancy) who are experiencing food insecurity (defined as a positive screening on the Hunger Vital Sign questionnaire) to receive nutritional support.

At MGH, the investigators have partnered with 3 Social Service Organizations (SSOs) to deliver 3 types of nutritional support. Community Servings provides medically tailored meals with nutritional counseling. Fresh Food Generation provides healthy food boxes. Fresh Connect provides debit cards with monthly allotments that can be used to purchase produce.

The current workflow for identifying and enrolling appropriate ACO members relies largely on referrals from Primary Care Teams. Role groups who respond to social needs within primary care, such as Community Health Workers, integrated Care Managers, Community Resource Navigators and Emergency Department Navigators (collectively herein referred to as Care Managers), have been trained on the program's eligibility requirements and encouraged to offer enrollment to the patients they are working with. However, this current method in inadequate to identify many eligible patients. Only a very small subset of patients (less than 10%) with social needs identified on their primary care screening questionnaire are referred to Care Managers. In addition, Care Managers do not have any consistent method for identifying patients and offering the Flex Nutrition Program.

For patients interested in enrollment, Care Managers refer to two dedicated FLEX staff. Upon receipt of a referral, these two staff complete a Verification, Planning and Referral (VPR) form in EPIC, which generates a referral for the appropriate SSO, who subsequently reaches out to enroll the patient.

The investigators seek to understand if proactive outreach to eligible patients increases enrollment into and utilization of the Medicaid ACO Flex Nutrition Program. To answer this question, the investigators will identify eligible members (patients in the Medicaid ACO with a positive food insecurity screening plus one or more defined health conditions, see Inclusion criteria for more details) via an EPIC Report and randomize them into 3 cohorts. Cohort A will receive high intensity proactive outreach via phone, Cohort B will receive low-intensity outreach via letter and Cohort C will receive usual care with no proactive outreach. The investigators will use an EPIC report to generate a list of eligible patients, defined as Adult and Pediatric patients cared for within MGH Primary Care in the Medicaid ACO with a health needs-based criteria and a positive screening for food insecurity. Patients already enrolled into the Flex Nutrition program will be excluded.

The rationale for randomization is that our 2 FLEX staff have limited bandwidth to proactively outreach to all eligible patients. Randomizing eligible patients will ensure their efforts are distributed fairly and also allow the investigators to evaluate the effectiveness of low intensity and high intensity outreach. The Flex Services Nutrition Program is incorporated into routine clinical care at MGH.

ELIGIBILITY:
Inclusion Criteria:

Has Medicaid ACO as primary health insurance, confirmed food insecurity (defined as a positive screen on the Hunger Vital Sign, which is conducted in routine care within primary care) AND one of the following:

1. a Complex Physical Health Need
2. a Behavioral Health Need
3. a High Risk Pregnancy or
4. Repeated ED use.

A Complex Physical Health Need is defined as having a diagnosis of one or more of the following:

1. Obesity (adults with BMI > 30, pediatrics with weight in 95-99 percentiles)
2. Diabetes
3. Hypertension
4. Chronic kidney disease or end stage renal disease
5. Chronic heart failure
6. Adult or pediatric cancer diagnosis
7. Malnutrition
8. Failure to thrive
9. Gastrointestinal disease (e.g. inflammatory bowel disease such as Crohn's or Ulcerative Colitis)
10. Asthma and two or more uncontrolled exacerbations per year
11. COPD and two or more exacerbations per year High cholesterol
12. HIV / AIDs
13. Vitamin D deficiency or receiving Vitamin D supplements

A Behavioral Health Need is defined as one or more of the following:

1. Major depressive disorder
2. Generalized anxiety disorder
3. Bipolar disorder
4. Schizophrenia
5. Mood disorder (pediatric)
6. Developmental disorders (e.g. autism)
7. Substance use disorders or
8. (for adults) an individual with PHQ-9 score or GAD-7 score of 10 or greater.

High Risk Pregnancy is defined as:

High risk pregnant individual with a diagnosis of:

1. hypertensive disorders of pregnancy
2. pregestational or gestational diabetes
3. a referral to or care with a Maternal Fetal Medicine specialist or
4. other high-risk, high-acuity diagnoses that can benefit from meeting an unmet social need

Repeated ED Use is defined as:

2+ ED visits in last 6 months or 4+ ED visits in last 12 months

Exclusion Criteria:

1. Language other than English, Arabic, Spanish, or Creole.
2. Language unknown
3. Age> 64.5 years (patients age out of the Medicaid ACO at 65, and this is a 6 month intervention)
4. Previous referral (already in database whether or not enrolled)
5. Invalid address (e.g. exclude address="NPA")
6. No phone number
7. Same address as another patient in report (randomly select 1 to retain)

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Referred to Flex Nutrition Program | 3 months after outreach is completed
  The percentage of patients in each study arm who are referred to the FLEX Nutrition program (VPR form completed and sent to the SSO)
Enrollment into the Flex Nutrition Program | 3 months after outreach is completed
  The percentage of patients in each study arm who are enrolled into the FLEX Nutrition program (Enrolled with the SSO). We will utilize SSO rosters of enrolled patients as our data source.
Enrollment in the Flex Nutrition Program by Vendor | 3 months after outreach is complete
  For patients enrolled into Flex Nutrition, the percentage breakdown by SSO vendor
  1. Community Servings
  2. Fresh Food Generation
  3. Fresh Connect We will utilize SSO rosters of enrolled patients as our data source.
Utilization of the Flex Nutrition Program | 3 months after outreach is complete
  The percentage of patients in each study arm who used the FLEX Nutrition program at least once Numerator: patients with any positive utilization 3 mths after outreach is complete
  1. Community Servings: received at least 1 delivery
  2. Fresh Food Generation: received at least delivery
  3. Fresh Connect: have charged their card at least once We will utilize SSO rosters of patients receiving services as our data source.

SECONDARY OUTCOMES:
Preventable ED visits | 12 months pre-outreach compared to 12 months after outreach is completed
  Number of ED visits that did not result in an admission 12 months pre-outreach compared to 12 months after outreach is completed
Avoidable Inpatient Hospitalizations | 12 months pre-outreach compared to 12 months after outreach is completed
  Unplanned inpatient hospitalizations 12 months pre-outreach compared to 12 months after outreach is completed
Outpatient no-show rate | 12 months pre-outreach compared to 12 months after outreach is completed
  No show rate during the 12 months pre-outreach period compared to 12 months after outreach is completed.
BMI for patients who are overweight/obese | 12 months pre-outreach compared to 12 months after outreach is completed
  Of patients with elevated BMI (defined as BMI>25 prior to outreach completed), change in pre-outreach BMI compared to 12 months after outreach is completed
  BMI change for each patient: BMI pre-outreach (use last chronological value prior to outreach completed, within 12 months) - BMI 12 months after outreach is completed (If multiple values, use last chronological value post outreach, within 12 months)
A1c for patients with Impaired Fasting Glucose/Diabetes | 12 months pre-outreach compared to 12 months after outreach is completed
  Of patients with IFG/Diabetes (defined as Diagnosis of IFG/DM AND/OR a1c > 5.7 prior to outreach completed), change in pre-outreach a1c compared to 12 months after outreach is completed.
  A1c change for each patient: a1c pre-outreach (If multiple values, use last chronological value prior to outreach completed, within 12 months) - a1c 12 months after outreach is completed (If multiple values, use last chronological value post outreach, within 12 months)
Blood Pressure for patients with HTN | 12 months pre-outreach compared to 12 months after outreach is completed
  Of patients with Hypertension (defined as Diagnosis of Hypertension AND/OR BP > 130/80 prior to outreach completed), change in pre-outreach Blood Pressure compared to 12 months after outreach is completed.
  BP change for each patient: BP 12 mths pre-outreach (If multiple values, take mean of all values. If more than 1 value on one day, take the lowest value measured on that day) - BP during 12 months post-outreach period (If multiple values, take mean of all values. If more than 1 value on one day, take the lowest value measured on that day.)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Matathia, MD MPH, Principal Investigator — MGH

IPD SHARING:
Plan to Share IPD: No